CLINICAL TRIAL: NCT01116427
Title: A Phase II, Randomized, Double-blind, Parallel-group, Placebo-controlled, Multicenter Study to Evaluate the Safety and Efficacy of Abatacept in Adults With Relapsing-remitting Multiple Sclerosis
Brief Title: A Cooperative Clinical Study of Abatacept in Multiple Sclerosis
Acronym: ACCLAIM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT ITN035AI
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Results first posted 2016-04-08 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: MS; multiple sclerosis; relapsing-remitting multiple sclerosis; RRMS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abatacept (Experimental): Receives abatacept during first course of treatment, switching to placebo during extension phase.
  Interventions: Biological: abatacept; Drug: Placebo
- Placebo, followed by abatacept (Placebo Comparator): Receives a placebo for first course of treatment, switching to abatacept in the extension phase.
  Interventions: Biological: abatacept; Drug: Placebo

INTERVENTIONS:
Biological: abatacept — In core/extension phase: administered IV at weeks 0/28, 2/30, and 4/32, and then every 4 weeks until week 24/52; Dosing: less than 60 kg, 500 mg; 60-100 kg, 750 mg; or greater than 100 kg, 1 gram
  Other Names: Orencia®; CTLA4-Ig
Drug: Placebo — In core/extension phase: administered IV at weeks 0/28, 2/30, and 4/32, and then every 4 weeks until week 24/52
  Other Names: placebo abatacept

SUMMARY:
The ACCLAIM study is testing whether the medication "abatacept" can be of benefit to patients with relapsing-remitting multiple sclerosis (MS). Although abatacept is an investigational medication for MS, it is not a new drug. Abatacept has been approved by the FDA to treat rheumatoid arthritis.

DETAILED DESCRIPTION:
MS is a chronic autoimmune disease in which blood cells that are supposed to protect the body from infection mistakenly attack the body's own tissue. In MS, the target of this attack is a protein called myelin that coats nerves throughout the body. Damage to this protective layer can lead to loss of neurologic function.

There are a number of treatments available to MS patients. Interferon beta, Copaxone, and other drugs can delay the worsening of the disease in some patients. For other patients, more aggressive treatment with chemotherapy drugs such as cyclophosphamide or azathioprine are needed. These drugs attempt to slow the disease by limiting the activity of the entire immune system. Because of this, they can often have serious side effects.

This study evaluates the efficacy of abatacept in the treatment of relapsing-remitting MS. In the first phase of the study, all participants will receive 8 intravenous treatments over a period of 24 weeks. Then, if a participant remains eligible, they will enter the second phase of the study and will receive another 8 treatments over the following 24 weeks. Two-thirds (2 out of 3) of participants will receive the study drug abatacept in the first phase, and then an inactive form (placebo) of the drug in the second phase. The remaining one-third (1 in 3) will get the placebo first, then the study drug in the second phase if they remain eligible. Therefore, all participants in the ACCLAIM trial will have the opportunity to receive the study drug abatacept if they remain healthy during the study. Participants will be asked to return for a follow-up visit 12 weeks after all treatments have been completed.

Regular appointments scheduled during the trial will be used to monitor participants' health and progress in the study. These appointments will include: physical and neurological exams, blood tests and motor function assessments. A total of 11 magnetic resonance imaging (MRI) procedures are scheduled during the study. The study medication and procedures related to the study will be provided at no expense to the participant.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite Relapsing-remitting Multiple Sclerosis (RRMS) meeting McDonald's criteria
* Expanded Disability Status Scale (EDSS) scores between 0 and 5
* Active disease as defined by at least one of the following criteria:

  1. One or more documented clinical exacerbations in the past year prior to visit -2
  2. One or more gadolinium (Gd)-enhanced MRI lesions in the past year
* Willingness to forego available MS therapies
* Ability and willingness to provide informed consent and comply with study requirements and procedures

Exclusion Criteria:

* Normal brain MRI at week -5 scan
* Females who are pregnant, intending pregnancy, or lactating, and unwilling to undergo pregnancy testing
* Females who are unwilling to use approved methods of contraception for the duration of the study
* Any chronic medical disease, other than MS, that compromises organ function
* Active infection
* Diagnosis of secondary or primary progressive MS
* Previous treatment with cyclophosphamide, mitoxantrone, cladribine, or rituximab at any time
* Previous treatment with abatacept within the last 52 weeks prior to visit -2
* Previous treatment with systemic steroids, interferon, Copaxone, mycophenolate, or other immunosuppressive medications within the last 4 weeks prior to visit -2
* Previous treatment with Natalizumab within the last 26 weeks prior to visit -2
* Previous vaccination with live vaccine, or previous treatment with fingolimod, within the last 8 weeks prior to visit-2
* Diagnosis of malignancy other than basal cell carcinoma or cervical carcinoma in situ
* Claustrophobia or other contraindications to Gd-enhanced MRI
* Positive for human immunodeficiency virus (HIV) serology
* Positive for hepatitis B surface antigen (HBsAg)
* Positive for hepatitis C virus (HCV) serology
* Purified protein derivative (PPD)-tuberculin skin test result greater than 5 mm induration
* Hemoglobin less than 10.5 gm/dL
* Platelets less than 100K/µL
* Absolute lymphocyte count less than 700 cells/μL
* Serum creatinine greater than 1.20 mg/dL
* eGFR (estimated glomerular filtration rate) less than 60 mL/min/1.73 m^2
* IgG anti-cardiolipin antibody greater than 15 GPL U/mL
* Previous participation in another interventional clinical trial within the past 4 weeks prior to visit -2
* Allergy or sensitivity to any component of abatacept
* The presence of any medical condition that the investigator deems incompatible with participation in the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-09; Primary Completion 2014-06 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samia Khoury, MD, Principal Investigator — Brigham and Women's Hospital
Locations (21):
- United States (20):
  - St. Josephs Hospital and Medical Center - Barrow Neurology, Phonix, Arizona
  - Jordan Research and Education Institute (REDI): Alta Bates Summit Medical Center, Berkeley, California
  - University of Southern California - Keck School of Medicine, Los Angeles, California
  - Newport Beach Clinical Research Associates, Inc., Newport Beach, California
  - University of California, Davis, Sacramento, California
  - University of Miami, Miami, Florida
  - South Suburban Neurology, Flossmoor, Illinois
  - Norton Neuroscience Institute - Norton Neurology Services MS Center, Louisville, Kentucky
  - Louisiana State University, Shreveport, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Judith Jaffe Multiple Sclerosis Center: Weill Cornell Medical College, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Neurology Specialists, Inc., Dayton, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The Neurology Foundation, Inc., Providence, Rhode Island
  - Advanced Neurosciences Institute, Franklin, Tennessee
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data in: 1.)ImmPort, a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts that also provides data analysis tools that are available to researchers who register online and subsequently receive DAIT approval; and 2.)TrialShare, a clinical trials research portal developed by the Immune Tolerance Network that makes data from the consortium's clinical trials publicly available without charge.

REFERENCES:
- [Background] Viglietta V, Bourcier K, Buckle GJ, Healy B, Weiner HL, Hafler DA, Egorova S, Guttmann CR, Rusche JR, Khoury SJ. CTLA4Ig treatment in patients with multiple sclerosis: an open-label, phase 1 clinical trial. Neurology. 2008 Sep 16;71(12):917-24. doi: 10.1212/01.wnl.0000325915.00112.61. PMID 18794494
- [Result] Khoury SJ, Rochon J, Ding L, Byron M, Ryker K, Tosta P, Gao W, Freedman MS, Arnold DL, Sayre PH, Smilek DE; ACCLAIM Study Group. ACCLAIM: A randomized trial of abatacept (CTLA4-Ig) for relapsing-remitting multiple sclerosis. Mult Scler. 2017 Apr;23(5):686-695. doi: 10.1177/1352458516662727. Epub 2016 Aug 5. PMID 27481207
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/Pages/default.aspx
- See also: Immune Tolerance Network (ITN) — http://www.immunetolerance.org
- See also: ITN TrialShare: open public access to study level information — http://www.itntrialshare.org
- Available data/document: Study protocol synopsis, -navigator, -schedule of assessments, study schema, and manuscript(s) with overviews, data and reports, participant level data: ACCLAIM ITN035AI — https://www.itntrialshare.org/project/Studies/ITN035AIPRI/Study%20Data/begin.view? — ACCLAIM ITN035AI is the Study Identifier in the Immune Tolerance Network (ITN) TrialShare Clinical Trials Research Portal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with relapsing-remitting multiple sclerosis were recruited from 21 sites in the US and Canada between November 2010 and November 2013
Groups:
- Abatacept First, Then Placebo: Subjects received abatacept intravenously (IV) at weeks 0, 2, and 4, and then every 4 weeks through week 24. After week 24, participants eligible for the extension phase of the trial received placebo IV on weeks 28, 30, and 32 then every 4 weeks until week 52. Participants completed an additional 12 weeks of observation until week 64. Dosing of abatacept was as follows:Participants weighing less than 60 kg received 500 mg; 60-100 kg received 750 mg; and greater than 100 kg received 1 g.
- Placebo First, Then Abatacept: Subjects received placebo IV at weeks 0, 2, and 4, and then every 4 weeks through week 24. After week 24, participants eligible for the extension phase of the trial received abatacept IV on weeks 28, 30, and 32 then every 4 weeks until week 52. Participants completed an additional 12 weeks of observation until week 64. Dosing of abatacept was as follows. Participants weighing less than 60 kg received 500 mg; 60-100 kg received 750 mg; and greater than 100 kg received 1 g.
Period: Core Phase
Arm/Group | Abatacept First, Then Placebo | Placebo First, Then Abatacept
Started | 44 | 21
Completed | 39 | 20
Not Completed | 5 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Worsening Multiple Sclerosis | 1 | 0
Period: Extension Phase
Arm/Group | Abatacept First, Then Placebo | Placebo First, Then Abatacept
Started | 38 (One participant that completed core phase did not meet eligibility for Extension Phase) | 20
Completed | 29 | 18
Not Completed | 9 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Not using appropriate birth control | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Abatacept First, Then Placebo: Subjects received abatacept IV at weeks 0, 2, and 4, and then every 4 weeks through week 24. After week 24, participants eligible for the extension phase of the trial received placebo IV on weeks 28, 30, and 32 then every 4 weeks until week 52. Participants completed an additional 12 weeks of observation until week 64. Dosing of abatacept was as follows: Participants weighing less than 60 kg received 500 mg; 60-100 kg received 750 mg; and greater than 100 kg received 1 g.
- Total: Total of all reporting groups
Arm/Group | Abatacept First, Then Placebo | Placebo First, Then Abatacept | Total
Number analyzed (Participants) | 44 | 21 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (9.7) | 42.7 (11.0) | 41.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 18 | 50
  Male | 12 | 3 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 41 | 20 | 61
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 35 | 16 | 51
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 41 | 19 | 60
  United States | 3 | 2 | 5
Baseline Expanded Disability Status Scale (EDSS) Score [Mean (Standard Deviation); unit: units on a scale] — Baseline EDSS score was the lowest score observed at either visit -2 (Wk -5) or visit -1 (Wk -1). The EDSS is an assessment for severity of multiple sclerosis. The EDSS an ordinal clinical rating scale ranging from 0 (normal neurological examination) to 10 (death due to multiple sclerosis) in half-point increments.
  units on a scale | 2.0 (1.3) | 2.4 (1.2) | 2.1 (1.3)
Baseline Multiple Sclerosis Functional Composite (MSFC) Score [Mean (Standard Deviation); unit: Scores on a scale] — Baseline MSFC score was the most recent score on or before Randomization. The three component measures of the MSFC include the 1) Time 25-foot Walk (a measure of lower extremity function), 2) 9-hole Peg Test (a measure of upper extremity function), and 3) Paced Auditory Serial Addition Test (a measure of cognitive function). Scores from all three components are combined then are converted into a Z-score for analyses, with a range from -1 to 1. A positive score indicates less severity of multiple sclerosis while negative scores indicate more severe multiple sclerosis symptoms.
  Scores on a scale | -0.01 (0.68) | 0.03 (0.81) | 0.00 (0.72)
Baseline Gd-enhanced Lesions [Mean (Standard Deviation); unit: Lesions] — Number of gadolinium (Gd)-enhancing lesions detected during an MRI scan. Baseline MRI evaluations were obtained at Visit -1 (Wk -1). Gd-enhancing lesions are measured on T1 weighted images after injection of 0.1 mM/kg of gadolinium pentate. A higher score indicates more severe multiple sclerosis.
  Lesions | 0.7 (1.4) | 3.8 (10.7) | 1.7 (6.3)
Baseline T2 Lesion Volume [Mean (Standard Deviation); unit: cm^3] — Total volume of all T2 lesions detected during an MRI scan. Baseline MRI evaluations were obtained at Visit -1 (Wk -1). A T2 lesion is defined as an abnormal, hyperintense white-matter area visible on T2 weighted images. A higher score indicates more severe multiple sclerosis.
  cm^3 | 6.7 (8.1) | 9.6 (9.0) | 7.7 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of New Inflammatory MRI Lesions Per Monthly Scans
Description: The mean number of new inflammatory MRI lesions obtained on scans every 4 weeks from Week 8 to Week 24, adjusted for differences between subjects before treatment by subtracting the number of new inflammatory lesions observed from the week -1 MRI scan . An inflammatory lesion is defined as a gadolinium (Gd)-enhancing lesion that shows hyperintensity on postcontrast but no hyperintensity on noncontrast T1 images. A new inflammatory lesion is one that was not present on the previously scheduled MRI scan. If the previously scheduled MRI scan was missing, the scan was compared to the last available MRI.
Time Frame: Weeks 8-24
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: New Lesions
Arm/Group | Abatacept First, Then Placebo | Placebo First, Then Abatacept
Number analyzed (Participants) | 42 | 20
New Lesions | 0.4 (0.9) | 1.7 (3.6)
Statistical Analysis 1: Comparison: Abatacept First, Then Placebo vs Placebo First, Then Abatacept; Test type: Superiority or Other; p = 0.87, Wilcoxon (Mann-Whitney) — Analysis was stratified on the presence or absence of subclinical activity as demonstrated by a Gd-enhanced lesion on one MRI in the past year prior to enrollment

2. Secondary Outcome: Absolute Number of New Inflammatory MRI Lesions on Monthly Scans
Description: The absolute number of new inflammatory MRI lesions obtained on scans every 4 weeks from Week 8 to Week 24. An inflammatory lesion is defined as a gadolinium (Gd)-enhancing lesion that shows hyperintensity on postcontrast but no hyperintensity on noncontrast T1 images. A new inflammatory lesion is one that was not present on the previously scheduled MRI scan. If the previously scheduled MRI scan was missing, the scan was compared to the last available MRI.
Time Frame: Weeks 4-24
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: New Lesions
Arm/Group | Abatacept First, Then Placebo | Placebo First, Then Abatacept
Number analyzed (Participants) | 42 | 20
New Lesions | 2.3 (4.1) | 9.1 (18.8)
Statistical Analysis 1: Comparison: Abatacept First, Then Placebo vs Placebo First, Then Abatacept; Test type: Superiority or Other; p = 0.36, Wilcoxon (Mann-Whitney) — Wilcoxon rank sum test in which the total number of new lesions were converted to ranks and then compared between groups

3. Secondary Outcome: Lesion Volume Accumulation on T2-weighted MRI Scans Over 24 Weeks
Description: Difference in total volume of all T2 lesions detected at Week 24 MRI scan compared to Week -1 MRI scan. A T2 lesion is defined as an abnormal, hyperintense white-matter area visible on T2 weighted images. A higher score indicates more severe multiple sclerosis.
Time Frame: Week -1 to Week 24
Population: Intent-to-treat population that did not terminate study prior to Week 24
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Abatacept First, Then Placebo | Placebo First, Then Abatacept
Number analyzed (Participants) | 39 | 19
cm^3 | -0.05 (0.42) | -0.18 (1.27)
Statistical Analysis 1: Comparison: Abatacept First, Then Placebo vs Placebo First, Then Abatacept; Test type: Superiority or Other; p = 0.93, Wilcoxon (Mann-Whitney) — Rank sum test in which the lesion volume change values per participant were converted to ranks and compared between the treatment groups

4. Secondary Outcome: Percent Brain Volume Change
Description: Percent Brain Volume Change is a measure of brain atrophy. Brain volume was calculated from a MRI scan at Week -1 and a MRI scan at Week 24 then the percent change from Week -1 to Week 24 was calculated. A negative change score means volume decreased. A decrease in volume indicates progression of multiple sclerosis severity.
Time Frame: Week -1 to Week 24
Population: Intent-to-treat population that did not terminate study prior to Week 24 and had MRI scans at both Week -1 and Week 24
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Abatacept First, Then Placebo | Placebo First, Then Abatacept
Number analyzed (Participants) | 39 | 18
percent change | -0.09 (0.54) | -0.25 (0.53)
Statistical Analysis 1: Comparison: Abatacept First, Then Placebo vs Placebo First, Then Abatacept; Test type: Superiority or Other; p = 0.68, Wilcoxon (Mann-Whitney) — Wilcoxon rank sum test in which percent brain volume change values per participant were converted to ranks and the ranks were compared between groups

5. Secondary Outcome: Mean Number of New Inflammatory Lesions in 8-week Intervals
Description: The mean number of new inflammatory MRI lesions obtained on scans every 8 weeks from Week 8 to Week 24. An inflammatory lesion is defined as a gadolinium (Gd)-enhancing lesion that shows hyperintensity on postcontrast but no hyperintensity on noncontrast T1 images. A new inflammatory lesion is one that was not present on the previously scheduled MRI scan. If the previously scheduled MRI scan was missing, the scan was compared to the last available MRI.
Time Frame: Week 8 to Week 24
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: New Lesions
Arm/Group | Abatacept First, Then Placebo | Placebo First, Then Abatacept
Number analyzed (Participants) | 42 | 20
New Lesions | 0.5 (1.2) | 2.2 (4.9)
Statistical Analysis 1: Comparison: Abatacept First, Then Placebo vs Placebo First, Then Abatacept; Test type: Superiority or Other; p = 0.21, Wilcoxon (Mann-Whitney) — Wilcoxon rank sum test in which mean numbers of new lesions per participant were converted to ranks and compared between groups

6. Secondary Outcome: Number of Participants Progressing on the EDSS Scale by at Least 1 Point
Description: The Expanded Disability Status Scale (EDSS) is an assessment for severity of multiple sclerosis. The EDSS an ordinal clinical rating scale ranging from 0 (normal neurological examination) to 10 (death due to multiple sclerosis) in half-point increments. Baseline EDSS score was the lowest score observed at either visit -2 (Wk -5) or visit -1 (Wk -1). EDSS progression is defined as an increase of at least 1 point on the EDSS compared to baseline if the baseline was greater than 1.0, or 1.5 points on EDSS if baseline was less than or equal to 1.0, which persisted for a minimum of 12 weeks or was found on three consecutive EDSS assessments starting at Visit 3 (Wk 8).
Time Frame: Week -1 to Week 24
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Abatacept First, Then Placebo | Placebo First, Then Abatacept
Number analyzed (Participants) | 42 | 20
participants | 5 | 1
Statistical Analysis 1: Comparison: Abatacept First, Then Placebo vs Placebo First, Then Abatacept; Test type: Superiority or Other; p = 0.65, Fisher Exact

7. Secondary Outcome: Annualized Relapse Rate
Description: The rate of multiple sclerosis relapse by year. Annualized relapse rate is calculated by dividing the total number of relapse events in the core phase in each treatment group by the total number of days participants participated in the study during the core phase. This number is then multiplied by 365.25 to get an annualized rate.
Time Frame: Week -1 to Week 24
Population: Intent-to-treat
Measure: Number; unit: Relapse Rate by Year
Arm/Group | Abatacept First, Then Placebo | Placebo First, Then Abatacept
Number analyzed (Participants) | 42 | 20
Relapse Rate by Year | 0.13 | 0.09

8. Secondary Outcome: Mean Change in the MSFC Over 24 Weeks of Treatment
Description: The Multiple Sclerosis Functional Composite (MSFC) is a three-part, standardized, quantitative assessment instrument to measure severity of multiple sclerosis. The MSFC combines three component measures to create a composite measure. The three component measures of the MSFC include the 1) Time 25-foot Walk (a measure of lower extremity function), 2) 9-hole Peg Test (a measure of upper extremity function), and 3) Paced Auditory Serial Addition Test (a measure of cognitive function). Mean change in MSFC scores from baseline to Week 24 were assessed. Scores from all three components are combined then are converted into a Z-score for analyses, with a range from -1 to 1. A positive score indicates improvement in the severity of multiple sclerosis symptoms while negative scores indicate decline in multiple sclerosis symptoms.
Time Frame: Week -1 to Week 24
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Abatacept First, Then Placebo | Placebo First, Then Abatacept
Number analyzed (Participants) | 42 | 20
Scores on a scale | 0.10 (0.30) | -0.04 (0.40)
Statistical Analysis 1: Comparison: Abatacept First, Then Placebo vs Placebo First, Then Abatacept; Test type: Superiority or Other; p = 0.13, Wilcoxon (Mann-Whitney) — Wilcoxon rank sum test in which the change from baseline scores per subject were converted to ranks and compared between treatment groups

9. Secondary Outcome: Mean Number of New Inflammatory MRI Lesions Per Scan During the Extension Phase
Description: The mean number of new inflammatory MRI lesions obtained on scans at Weeks 36 and 52, adjusted for differences between subjects before treatment by subtracting the number of new inflammatory lesions observed from the week 24 MRI scan. An inflammatory lesion is defined as a gadolinium (Gd)-enhancing lesion that shows hyperintensity on postcontrast but no hyperintensity on noncontrast T1 images. A new inflammatory lesion is one that was not present on the previously scheduled MRI scan. If the previously scheduled MRI scan was missing, the scan was compared to the last available MRI.
Time Frame: Weeks 36 and 52
Population: Intent-to-treat in Extension Phase
Measure: Mean (Standard Deviation); unit: New Lesions
Arm/Group | Abatacept First, Then Placebo | Placebo First, Then Abatacept
Number analyzed (Participants) | 34 | 19
New Lesions | 1.3 (2.7) | 0.6 (1.0)
Statistical Analysis 1: Comparison: Abatacept First, Then Placebo vs Placebo First, Then Abatacept; Test type: Superiority or Other; p = 0.06, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

10. Secondary Outcome: Lesion Volume Accumulation on T2-Weighted MRI Scans Between 24 Weeks and 52 Weeks
Description: Difference in total volume of all T2 lesions detected at Week 52 MRI scan compared to Week 24 MRI scan. A T2 lesion is defined as an abnormal, hyperintense white-matter area visible on T2 weighted images. A higher score indicates more severe multiple sclerosis.
Time Frame: Week 24 to Week 52
Population: Intent-to-treat in Extension Phase who had an MRI at Week 52
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Abatacept First, Then Placebo | Placebo First, Then Abatacept
Number analyzed (Participants) | 26 | 16
cm^3 | 0.47 (0.99) | 0.07 (1.19)
Statistical Analysis 1: Comparison: Abatacept First, Then Placebo vs Placebo First, Then Abatacept; Test type: Superiority or Other; p = 0.07, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 3, analysis 1]

11. Secondary Outcome: Percent Brain Volume Change Between 24 Weeks and 52 Weeks
Description: Percent Brain Volume Change is a measure of brain atrophy. Brain volume was calculated from a MRI scan at Week 24 and a MRI scan at Week 25 then the percent change from Week 24 to Week 52 was calculated. A negative change score means volume decreased. A decrease in volume indicates progression of multiple sclerosis severity.
Time Frame: Week 24 to Week 52
Population: Intent-to-treat in Extension Phase who had an MRI at Week 52 with data to contribute to brain volume measurements
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Abatacept First, Then Placebo | Placebo First, Then Abatacept
Number analyzed (Participants) | 24 | 16
Percent change | -0.28 (0.42) | -0.31 (0.35)
Statistical Analysis 1: Comparison: Abatacept First, Then Placebo vs Placebo First, Then Abatacept; Test type: Superiority or Other; p = 0.88, Wilcoxon (Mann-Whitney) — Wilcoxon rank sum test in which the percent brain volume change values per participant were converted to ranks and compared between treatment groups

12. Secondary Outcome: Number of Participants Progressing on the EDSS Scale by at Least 1 Point
Description: The Expanded Disability Status Scale (EDSS) is an assessment for severity of multiple sclerosis. The EDSS an ordinal clinical rating scale ranging from 0 (normal neurological examination) to 10 (death due to multiple sclerosis) in half-point increments. Extension baseline EDSS score was the most recent non-missing value on or before Week 28. Only participants who scored between a 0 and a 5 at baseline were analyzed for this outcome measure. EDSS progression is defined as an increase of at least 1 point on the EDSS compared to baseline if the baseline was greater than 1.0, or 1.5 points on EDSS if baseline was less than or equal to 1.0, which persisted for a minimum of 12 weeks or was found on three consecutive EDSS assessments starting at Visit 3 (Wk 8).
Time Frame: Week 24 to Week 64
Population: Intent-to-treat in Extension Phase
Measure: Number; unit: participants
Arm/Group | Abatacept First, Then Placebo | Placebo First, Then Abatacept
Number analyzed (Participants) | 34 | 19
participants | 1 | 2
Statistical Analysis 1: Comparison: Abatacept First, Then Placebo vs Placebo First, Then Abatacept; Test type: Superiority or Other; p = 0.29, Fisher Exact

13. Secondary Outcome: Annualized Relapse in Extension Phase
Description: The rate of multiple sclerosis relapse by year. Annualized relapse rate is calculated by dividing the total number of relapse events in the extension and follow-up phases in each treatment group by the total number of days participants participated in the study during the extension and follow-up phases. This number is then multiplied by 365.25 to get an annualized rate.
Time Frame: Week 24 to Week 64
Population: Intent-to-treat in Extension Phase
Measure: Number; unit: Relapse Rate by Year
Arm/Group | Abatacept First, Then Placebo | Placebo First, Then Abatacept
Number analyzed (Participants) | 34 | 19
Relapse Rate by Year | 0.38 | 0.16

14. Secondary Outcome: Mean Change in the MSFC in Extension Phase
Description: The Multiple Sclerosis Functional Composite (MSFC) is a three-part, standardized, quantitative assessment instrument to measure severity of multiple sclerosis. The MSFC combines three component measures to create a composite measure. The three component measures of the MSFC include the 1) Time 25-foot Walk (a measure of lower extremity function), 2) 9-hole Peg Test (a measure of upper extremity function), and 3) Paced Auditory Serial Addition Test (a measure of cognitive function). Mean change in MSFC scores from Week 24 to Week 52 were assessed. Scores from all three components are combined then are converted into a Z-score for analyses, with a range from -1 to 1. A positive score indicates improvement in the severity of multiple sclerosis symptoms while negative scores indicate decline in multiple sclerosis symptoms.
Time Frame: Week 24 to Week 52
Population: Intent-to-treat in Extension Phase who Completed the MSFC at Week 52
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Abatacept First, Then Placebo | Placebo First, Then Abatacept
Number analyzed (Participants) | 27 | 18
Scores on a scale | 0.06 (0.21) | -0.01 (0.46)
Statistical Analysis 1: Comparison: Abatacept First, Then Placebo vs Placebo First, Then Abatacept; Test type: Superiority or Other; p = 0.67, Wilcoxon (Mann-Whitney) — Wilcoxon rank sum test in which the change from baseline scores per participant were converted to ranks and compared between treatment groups

ADVERSE EVENTS:
Time Frame: From enrollment until end of study (up to 64 weeks).
Description: Participants At Risk:1.) for the Core Phase=all who received at least one dose in the Core Phase 2.) for the Extension Phase=all who received at least one dose in the Extension Phase; and 3.) for the Follow-up Phase =all participants who completed the Extension Phase.
Groups:
- Core Phase: Abatacept -> Placebo: Subjects received abatacept intravenously (IV) at weeks 0, 2, and 4, and then every 4 weeks through week 24. Dosing of abatacept was as follows:
  Participants weighing-
  * less than 60 kg received 500 mg;
  * 60-100 kg received 750 mg; and
  * greater than 100 kg received 1 g.
- Core Phase: Placebo -> Abatacept: Subjects received placebo IV at weeks 0, 2, and 4, and then every 4 weeks through week 24.
- Extension Phase: Abatacept -> Placebo: After week 24, participants in Abatacept -> Placebo group eligible for the extension phase of the trial received placebo IV on weeks 28, 30, and 32 then every 4 weeks until week 52.
- Extension Phase: Placebo -> Abatacept: After week 24, participants in the Placebo -> Abatacept group eligible for the extension phase of the trial received abatacept IV on weeks 28, 30, and 32 then every 4 weeks until week 52. Dosing of abatacept was as follows:
  Participants weighing-
  * less than 60 kg received 500 mg;
  * 60-100 kg received 750 mg; and
  * greater than 100 kg received 1 g.
- Follow-up Phase: Abatacept -> Placebo: Following Week 52, participants in the Abatacept -> Placebo group completed an additional 12 weeks of observation until week 64.
- Follow-up Phase: Placebo -> Abatacept: Following Week 52, participants in the Placebo -> Abatacept group completed an additional 12 weeks of observation until week 64.
Arm/Group | Core Phase: Abatacept -> Placebo | Core Phase: Placebo -> Abatacept | Extension Phase: Abatacept -> Placebo | Extension Phase: Placebo -> Abatacept | Follow-up Phase: Abatacept -> Placebo | Follow-up Phase: Placebo -> Abatacept
Serious Adverse Events (participants affected / at risk) | 2/44 | 0/21 | 2/37 | 0/19 | 4/29 | 1/18
Other Adverse Events (participants affected / at risk) | 23/44 | 14/21 | 17/37 | 15/19 | 1/29 | 3/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Phase: Abatacept -> Placebo (N=44) | Core Phase: Placebo -> Abatacept (N=21) | Extension Phase: Abatacept -> Placebo (N=37) | Extension Phase: Placebo -> Abatacept (N=19) | Follow-up Phase: Abatacept -> Placebo (N=29) | Follow-up Phase: Placebo -> Abatacept (N=18)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster ophthalmic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Phase: Abatacept -> Placebo (N=44) | Core Phase: Placebo -> Abatacept (N=21) | Extension Phase: Abatacept -> Placebo (N=37) | Extension Phase: Placebo -> Abatacept (N=19) | Follow-up Phase: Abatacept -> Placebo (N=29) | Follow-up Phase: Placebo -> Abatacept (N=18)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (5) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (5) | 3 (5) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mean cell haemoglobin concentration decreased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (11) | 4 (5) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 3 (4) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Muscle spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No